CLINICAL TRIAL: NCT00070343
Title: Continuation Protocol For G3139 (Bcl-2 Antisense Oligonucleotide) And Dacarbazine In Patients With Malignant Melanoma Who Responded To This Combination In Protocol GM301
Brief Title: Oblimersen and Dacarbazine in Treating Patients With Advanced Malignant Melanoma That Has Responded to Treatment on Clinical Trial GENTA-GM301
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000331927; UCLA-0307016; GENTA-GM214
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2004-11

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; stage III melanoma
MeSH Terms: conditions — Melanoma | interventions — oblimersen; Dacarbazine

INTERVENTIONS:
Biological: oblimersen sodium
Drug: dacarbazine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as dacarbazine, use different ways to stop tumor cells from dividing so they stop growing or die. Oblimersen may help dacarbazine kill more tumor cells by making them more sensitive to the drug.

PURPOSE: This clinical trial is studying how well giving oblimersen together with dacarbazine works in treating patients with advanced malignant melanoma that previously responded to treatment with oblimersen and dacarbazine on clinical trial GENTA-GM301.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Provide continuation therapy with oblimersen (G3139) and dacarbazine to patients with advanced malignant melanoma who obtained response or stabilization of disease after prior treatment with this therapy on GENTA-GM301.

Secondary

* Determine serious adverse events in patients treated with this regimen.

OUTLINE: This is a nonrandomized, open-label, multicenter, continuation study.

Patients receive oblimersen (G3139) IV continuously on days 1-5 and dacarbazine IV over 1 hour on day 5. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients who complete 8 courses of treatment may receive additional courses at the discretion of the physician.

Patients are followed every 2 months for up to 2 years after initiation of GENTA-GM301 protocol.

PROJECTED ACCRUAL: A total of 375 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced malignant melanoma

  * Unresectable or metastatic disease
* Previously enrolled on GENTA-GM301 protocol

  * Complete or partial objective response or stable disease after completion of 8 courses of oblimersen (G3139) and dacarbazine on arm II of GENTA-GM301
* Measurable or evaluable disease
* No uncontrolled brain metastases or leptomeningeal disease

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3*
* Platelet count at least 100,000/mm^3*
* Hemoglobin at least 8 g/dL* NOTE: *Hematopoietic growth factor or transfusion independent

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Albumin at least 2.5 g/dL
* PTT no greater than 1.5 times ULN
* PT no greater than 1.5 times ULN OR
* INR no greater than 1.3
* No history of chronic hepatitis or cirrhosis

Renal

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 50 mL/min

Cardiovascular

* No uncontrolled congestive heart failure
* No active symptoms of coronary artery disease, defined as uncontrolled arrhythmias or recurrent chest pain despite prophylactic medication
* No New York Heart Association class III or IV heart disease
* No cardiovascular signs and symptoms grade 2 or greater within the past 4 weeks

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other significant medical disease
* No uncontrolled seizure disorder
* No active infection
* No uncontrolled diabetes mellitus
* No active autoimmune disease
* No known hypersensitivity to phosphorothioate-containing oligonucleotides or dacarbazine
* No intolerance to prior oblimersen and dacarbazine, including discontinuation of protocol therapy due to 1 or more adverse events
* HIV negative
* Satisfactory venous access for a 5-day continuous infusion
* Intellectually, emotionally, and physically able to maintain an ambulatory infusion pump

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior biologic therapy, immunotherapy, cytokine therapy, or vaccine therapy and recovered
* No concurrent anticancer biologic therapy

Chemotherapy

* See Disease Characteristics
* No other concurrent anticancer chemotherapy

Endocrine therapy

* No concurrent chronic corticosteroids (average dose of at least 20 mg/day of prednisone or equivalent)

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent anticancer radiotherapy

Surgery

* At least 4 weeks since prior major surgery and recovered

Other

* At least 4 weeks since other prior therapy and recovered
* More than 3 weeks since prior experimental therapy (except for GENTA-GM301 protocol)
* No intervening systemic therapy for melanoma since completion of GENTA-GM301 protocol therapy
* No other concurrent anticancer therapy, including investigational therapy
* No concurrent immunosuppressive drugs
* No concurrent anticoagulation therapy

  * Concurrent warfarin (1 mg/day) for central line prophylaxis is allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: John A. Glaspy, MD, MPH, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States